CLINICAL TRIAL: NCT05496933
Title: Colombia National Porphyria Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación Grupo de Investigación en Cuidados Intensivos y Obstetricia (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Principal Investigator, José Antonio Rojas Suarez, Principal Investigator, Fundación Grupo de Investigación en Cuidados Intensivos y Obstetricia
Other Study IDs: 0112-2020
Record Dates: First submitted 2021-11-10; First posted 2022-08-11 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Rare Diseases; Porphyrias
Keywords: Acute Hepatic Porphyria; Porphyrias; Quality of life
MeSH Terms: conditions — Rare Diseases; Porphyrias; Coproporphyria, Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
porphyria is classified as a rare disease and is produced by defects in the enzymatic activity in the biosynthesis of the heme group that leads to the over-accumulation and excretion of porphyrin precursors in hepatocytes or erythroid cells, extrahepatic or extramedullary cells, tissue, and end-organ injury. Acute intermittent porphyria is the most common and severe form of hepatic porphyria, with an annual incidence of symptomatic patients of 0.13 per million people. Aim: characterization of cases of acute hepatic porphyria in Colombia. Methods: a descriptive pilot study of patients diagnosed with acute hepatic porphyria's in Colombia. Patients of all age groups with a confirmed diagnosis of acute hepatic porphyria. Patients with concomitant pathologies, as well as pregnant women, will also be included. Patients who refuse to participate in the study will be excluded. Expected results: describe the sociodemographic and clinical characteristics of patients with a diagnosis of acute hepatic porphyria, and encourage patients and/or representatives in the research agenda.

DETAILED DESCRIPTION:
A cross-sectional descriptive observational study is carried out in adult patients diagnosed with HAP in Colombia, the incidence and prevalence were estimated, the clinical, socio-demographic and acute attack characteristics are described, and the health-related quality of life was evaluated with the SF-36 questionnaire.

ELIGIBILITY:
Inclusion Criteria: - Patients of all age groups with a confirmed diagnosis of acute hepatic porphyria with AT LEAST ONE OF THE FOLLOWING CHARACTERISTICS will be included:

* Acute symptoms consistent with disease and positive urine qualitative porphobilinogen or substantially elevated quantitative porphobilinogen.
* Acute symptoms compatible with the disease and decreased HMBS enzyme activity (less than 50%).
* Mutation in the genetic sequence of the HMBS gene.
* Confirmatory test that identifies the type of porphyria (analysis of total and fractionated porphyrins in urine, feces and plasma).

Patients with concomitant pathologies, as well as pregnant women, will also be included.

Exclusion criteria:

* Patients who refuse to participate in the study will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria: - Patients of all age groups with a confirmed diagnosis of acute hepatic porphyria with AT LEAST ONE OF THE FOLLOWING CHARACTERISTICS will be included:
  * Acute symptoms consistent with disease and positive urine qualitative porphobilinogen or substantially elevated quantitative porphobilinogen.
  * Acute symptoms compatible with the disease and decreased HMBS enzyme activity (less than 50%).
  * Mutation in the genetic sequence of the HMBS gene.
  * Confirmatory test that identifies the type of porphyria (analysis of total and fractionated porphyrins in urine, feces and plasma).
  Patients with concomitant pathologies, as well as pregnant women, will also be included.
  Exclusion criteria:
  * Patients who refuse to participate in the study will be excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence | through study completion, an average of 3 year
  Total new cases of acute porphyry
Prevalence | through study completion, an average of 3 year
  Total cases of acute porphyry in Colombia
Life quality | through study completion, an average of 3 year
  Describe the well-being of patients, seeks to measure the impact that medical interventions have on the level of well-being of the patient, limiting itself to the experience that he has of his illness and its impact on it, evaluated with the The Short Form Health Survey 36 (SF-36 questionnaire: there are 36 questions, the possible score is from 0 to 100, with a higher score indicating a better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Gestion Salud, Cartagena, Departamento de Bolívar, Colombia